CLINICAL TRIAL: NCT02195336
Title: Diffusion MR (dMRT) During First Line Treatment of Non Squamous Lung Cancer With Chemotherapy Combined With Bevacizumab: Time Course and Prognostic and Predictive Impact.
Brief Title: dMR During First Line Treatment of Non Squamous Lung Cancer: Time Course and Prognostic and Predictive Impact.
Acronym: BevMar
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Karl Kölbeck (Other)
Responsible Party: Sponsor-Investigator, Karl Kölbeck, MD, Consultant, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BevMar; ML29273 (Other: Karolinska)
Record Dates: First submitted 2014-07-14; First posted 2014-07-21 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2014-07

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- dMRT, Bevacizumab, Chemotherapy (Experimental): dMRT: Magnetic Resonance Tomograph, Baseline, day 8, day 28, day 92, progression/relapse.
  Bevacizumab: 7.5mg/kg every 3 weeks for 3 cycles. Standard of care NSCLC first-line chemotherapy, doublets containing paclitaxel and carboplatin are preferred, every 3 weeks for 3 cycles.
  Thereafter Bevacizumab 7.5mg/kg every 3 weeks until progression/relapse or unacceptable toxicity.
  Interventions: Device: dMRT; Drug: Bevacizumab; Drug: paclitaxel and carboplatin

INTERVENTIONS:
Device: dMRT — Baseline, day 8, day 28, day 92, progression/relapse.
  Other Names: Magnetic Resonance Tomograph
Drug: Bevacizumab — 7.5mg/kg every 3 weeks for 3 cycles. Thereafter every 3 weeks until progression/relapse or unacceptable toxicity.
  Other Names: Avastin
Drug: paclitaxel and carboplatin — Standard of care NSCLC first-line chemotherapy Every 3 weeks for 3 cycles. Doublets containing paclitaxel and carboplatin are preferred

SUMMARY:
To date, there are no methods to reliably select which patients with non-squamous non-small cell lung cancer (NSCLC) that benefit most from treatment with bevacizumab. Data have shown that high levels of plasma VEGF are prognostic and correlates with a worse disease outcome in some tumour types, including advanced NSCLC.

Recent data are suggestive of a predictive value of imaging techniques for early detection of antiangiogenic treatment efficacy in different cancers. To our knowledge there are no presented data available on correlation between changes in diffusion-weighted MR and response to bevacizumab treatment in lung cancer. The current study is designed as a pilot study to prospectively investigate changes in MR variables during treatment with bevacizumab and to detect signals of prognostic and/or predictive value of MR changes during treatment.

DETAILED DESCRIPTION:
A Non Interventional, open-label, single arm, single institution pilot study. Eligible patients will be monitored by diffusion-weighted magnetic resonance tomography (dMRT) during treatment with bevacizumab + chemotherapy for up to four cycles followed by bevacizumab maintenance therapy until disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained prior to any study-specific procedure
2. Age ≥18 years
3. Able to comply with the protocol
4. Histologically or cytologically documented inoperable, metastatic (Stage IV) non small cell lung cancer
5. ECOG PS status 0-1
6. Life expectancy ≥12 weeks
7. Adequate haematological function:

   * Normal values of absolute neutrophil and platelet count, and a hemoglobin value ≥9 g/dL
8. Adequate liver function:

   * Total bilirubin <1.5 x ULN, AST, ALT <2.5 x ULN
9. Adequate renal function:

   * Calculated creatinine clearance ≥50 mL/min, a urine dipstick for proteinuria <2+.
10. Normal values of INR within 7 days prior to enrolment
11. If female, should not be pregnant or breast-feeding. Women with an intact uterus (unless amenorrhoeic for the last 24 months) must have a negative serum pregnancy test within 28 days prior to enrolment into the study.

Exclusion Criteria:

1. Mixed, non-small cell and small cell tumours or mixed adenosquamous carcinomas with a predominant squamous component
2. Known EGFR mutation or ALK translocation
3. History of haemoptysis
4. Evidence of tumour invading major blood vessels on imaging. The investigator or the local radiologist must exclude evidence of tumour that is fully contiguous with, surrounding, or extending into the lumen of a major blood vessel (e.g. pulmonary artery or superior vena cava)
5. Evidence of CNS metastases, even if previously treated. If suspected, the patient should be scanned within 28 days prior to enrolment to rule out CNS metastases
6. Previous treatment with chemotherapy or other anticancer agent
7. Previous radiotherapy of the primary tumour. Palliative extrathoracic radiotherapy is allowed prior to enrolment or during treatment
8. Major surgery (including open biopsy), significant traumatic injury within 28 days prior to enrolment or anticipation of the need for major surgery during study treatment
9. Minor surgery, including insertion of an indwelling catheter, within 24 hours prior to the first bevacizumab infusion
10. Current or recent (within 10 days of first dose of bevacizumab) use of aspirin (> 325mg/day) or use of full-dose oral or parenteral anticoagulants or thrombolytic agent for therapeutic purposes.
11. History or evidence of inherited bleeding diathesis or coagulopathy with the risk of bleeding
12. Uncontrolled hypertension (systolic >150 mmHg and/or diastolic >100 mmHg)
13. Clinically significant (i.e. active) cardiovascular disease
14. Non-healing wound, active peptic ulcer or bone fracture
15. History of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 6 months of enrolment
16. Women with an intact uterus (unless amenorrhoeic for the last 24 months) not using effective, means of contraception during the study and for a period of 6 months following the last administration of bevacizumab. Men who do not agree to use effective contraception during the study and for a period of 90 days following the last administration of bevacizumab. Men who do not agree to use effective contraception during the study and for a period of 90 days following the last administration of bevacizumab
17. Treatment with any other investigational agent, or participation in another clinical trial within 28 days prior to enrolment
18. Known hypersensitivity to bevacizumab or any of its excipients, and any of the chemotherapies
19. Evidence of ongoing or active infection, any other disease, neurological or metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or puts the patient at high risk for treatment-related complications
20. Patients diagnosed with a tracheo-oesophageal fistula
21. History of thrombotic disorders within the last 6 months prior to enrolment.
22. Contraindications for MRI: pacemaker and/or non-MRI compatible metallic implants/objects/devices/fragments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
dMRT changes during treatment | Baseline, Day 8, Day 28, Day 92, At relapse.
  Diffusion magnetic resonance tomography of lung lesions.

SECONDARY OUTCOMES:
Response to treatment | Baseline, Day 92, at 5, 7, 9, 12, 15, 18, 24 mo during follow up
  CT of lungs, clinical examinations
3. Time to disease progression (defined as the time period from the start of first-line therapy to investigator assessed disease progression) | Baseline, Day 92, at 5, 7, 9, 12, 15, 18, 24 mo during follow up
  CT, clinical examinations
Duration of survival | At 5, 7, 9, 12, 15, 18, 24, 36 and 48 mo during follow up
  Defined as the time period from the start of first-line therapy to death.

CONTACTS AND LOCATIONS:
Overall Officials: Karl-Gustav Kölbeck, MD, Principal Investigator — Karolinska University Hospital, Dept of Lung and Allergy
Locations (1):
- Dept of Lung and Allergy, Karolinska university hospital, Stockholm, Sweden